CLINICAL TRIAL: NCT04397666
Title: RT-PCR on Conjunctival Sample for the Detection of SARS-Cov-2 in Patients With Covid-19
Acronym: P20/09
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Edouard KOCH, coordonator investigator, Versailles Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P20/09_COVEYES
Record Dates: First submitted 2020-05-20; First posted 2020-05-21 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: SARS-CoV Infection; Pinkeye
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Conjunctivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental)
  Interventions: Diagnostic Test: conjunctival RT PCR

INTERVENTIONS:
Diagnostic Test: conjunctival RT PCR — conjunctival sample in covid-19 patients

SUMMARY:
the purpose of the study is to study the detection of SARS-Cov-2 virus in the conjunctiva of covid-19 patients and the presence or absence of conjunctivitis in these patients

ELIGIBILITY:
Inclusion Criteria:

* Men and Women positive for SARS-Cov-2 on a RT-PCR test of a sample of respiratory airway
* Persons over 18 years of age
* patients of both sexes
* Member of a social security scheme
* Having signed the consent form

Exclusion Criteria:

* Minors not emancipated, persons out of state to express their consent
* Participation in intervention research on Covid-19 involving experimental treatment
* History of chronic disease conjunctiva
* Patient with one of the one of the criteria of following gravity:

  1. EN > or =30/min,
  2. Pao2/Fio2 = or < 300,
  3. confusion and/or disorientation,
  4. hypotension (Tas90mmhg, requiring aggressive filling),
  5. need for a invasive ventilation,
  6. septic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
the SARS-Cov-2 positivity rate in patients with Covid-19 with or without signs of conjunctivitis | 3 months
  to assess the SARS-Cov-2 positivity rate in patients with Covid-19 with or without signs of conjunctivitis

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de versailles, Le Chesnay, France

IPD SHARING:
Plan to Share IPD: Undecided